CLINICAL TRIAL: NCT03020277
Title: Use of a Smartphone© Application to Study Autism Spectrum Disorders (ASD)
Acronym: SMARTAUTISM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: Institut de Recherche en Santé Publique, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC16_0185
Record Dates: First submitted 2016-12-19; First posted 2017-01-13 (Estimated); Last update posted 2024-03-20 (Actual); Status verified 2024-01

CONDITIONS: Autism Spectrum Disorders
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Ecological Momentary Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ASD children families (Other)
  Interventions: Other: Ecological Momentary Assessment with Smartphone© Application

INTERVENTIONS:
Other: Ecological Momentary Assessment with Smartphone© Application — Filling of the application every 3 days for 6 months by subjects (parents of patients with ASD)

SUMMARY:
This is a prospective, longitudinal, exploratory, open study with a 6-month follow-up period to explore via a specific Smartphone© application the evolution of a child's behavior over 6 months and the (psychological and social) effects of these changes on the family.

DETAILED DESCRIPTION:
This is a prospective, longitudinal, exploratory, open study with a 6-month follow-up period to assess the feasibility of using a Smartphone© application designed for parents of patients with ASD and to longitudinally collect data on the quality of life and anxiety of parents of children with ASD and the children's functional symptoms over multiple weeks under natural conditions.

Population:

The investigators propose to study individuals diagnosed with ASD based on National Health Authority (HAS) recommendations (on ADI-R diagnoses) from 3-16 years of age in the Pays de la Loire region. The investigators propose to include 100 families. The study is exploratory in nature; thus, randomizing patients is unnecessary. The investigators will include the first 100 families agreeing to participate in the study and meeting the inclusion criteria. All participants will be recruited from the Department of Child and Adolescent Psychiatry of University Hospital of Nantes and from the Regional Center for Autism (CRA des Pays de la Loire).

Method:

At the inclusion visit, parents will receive a code to download the app from the "application store" of their choice (depending on their Smartphone©) and sign an informed consent form.

All type 1 data from the inclusion visit will be stored in an electronic database and in the Smartphone© application (during the setup process).

This initial evaluation by the investigator will include the following type 1 data:

* Sibling rank and marital status,
* Lifestyle: rural or urban; single or multiple occupants of the chid's bedroom and housing type and surface,
* Educational and teaching load and conditions (special education, inclusive education, partial or full time, etc.), and
* The therapeutic management (speech therapy, psychomotor therapy, etc.).

Type 2 data will be stored in the electronic database only:

* Age at diagnosis,
* Current drug treatments (name, starting date and dose),
* Comorbidities (associated epilepsy, mental retardation and organic pathology),
* Medical and psychiatric family antecedent (ATCD),
* Original scores on the Autism Diagnostic Interview-Revised (ADI-R) and Autism Diagnostic Observation Schedule (ADOS) at the time of diagnosis, and
* Scores on the French version of the Childhood Autism Rating Scale (CARS) (http://www.autisme.qc.ca) at baseline and at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Having a child with an ASD diagnosis based on the International Classification of Diseases (ICD) 10 criteria.
* Having at least one Smartphone© (iOS Apple or Android).
* Signing the consent form for participation.

Exclusion Criteria:

* Having several children with an ASD diagnosis.
* Having children living in more than two areas

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2019-06-03 (Actual); Study Completion 2019-06-03 (Actual)

PRIMARY OUTCOMES:
Filling rate of the application | 6 months
  The primary outcome measure will be the filling rate (R) and the use of our application by the parents over six months. This number will be Automatically Generated by Application (AGA)
  Number of fillings = R 60

SECONDARY OUTCOMES:
child behavior with pairs | every 3 days for 6 months
  Secondary outcome measure include data from the application, that will be also Automatically Generated by the Application, which is filled by the parents, predominantly using a VAS from 0 (no) to 10 (severe) to measure the following variables
child sleep disorders | every 3 days for 6 months
  Secondary outcome measure include data from the application, that will be also Automatically Generated by the Application, which is filled by the parents, predominantly using a VAS from 0 (no) to 10 (severe) to measure the following variables
child eating disorders | every 3 days for 6 months
  Secondary outcome measure include data from the application, that will be also Automatically Generated by the Application, which is filled by the parents, predominantly using a VAS from 0 (no) to 10 (severe) to measure the following variables
child general behavior | every 3 days for 6 months
  Secondary outcome measure include data from the application, that will be also Automatically Generated by the Application, which is filled by the parents, predominantly using a Visual Analogic scale (VAS) from 0 (no) to 10 (severe) to measure the following variables
Visual Analogic scale quotation about parental self esteem | every 3 days for 6 months
  Visual Analogic scale (1 is bad to 10 is perfect ) quotation about parental self esteem by participants as assessed by SMARTAUTISM Application V1 2017 (Registered App)
Visual Analogic scale quotation about parental anxiety | every 3 days for 6 months
  Visual Analogic scale (1 is bad to 10 is perfect) quotation about parental anxiety by participants as assessed by SMARTAUTISM Application V1 2017 (Registered App)
Visual Analogic scale quotation about parental sleep | every 3 days for 6 months
  Visual Analogic scale (1 is bad to 10 is perfect) quotation about parental sleep by participants as assessed by SMARTAUTISM Application V1 2017 (Registered App)
Visual Analogic scale quotation about parental mood | every 3 days for 6 months
  Visual Analogic scale (1 is bad to 10 is perfect) quotation about parental mood by participants as assessed by SMARTAUTISM Application V1 2017 (Registered App)
Visual Analogic scale quotation about parental stress | every 3 days for 6 months
  Visual Analogic scale (1 is bad to 10 is perfect) quotation about parental stress by participants as assessed by SMARTAUTISM Application V1 2017 (Registered App)
Visual Analogic scale quotation about parental pain | every 3 days for 6 months
  Visual Analogic scale (1 is bad to 10 is perfect) quotation about parental pain by participants as assessed by SMARTAUTISM Application V1 2017 (Registered App)
Visual Analogic scale quotation about parental professional life | every 3 days for 6 months
  Visual Analogic scale (1 is unsatisfactory to 10 is satisfactory) quotation about parental professional life by participants as assessed by SMARTAUTISM Application V1 2017 (Registered App)
Visual Analogic scale quotation about parental personal life | every 3 days for 6 months
  Visual Analogic scale (1 is unsatisfactory to 10 is satisfactory) quotation about parental personal life by participants as assessed by SMARTAUTISM Application V1 2017 (Registered App)
Visual Analogic scale quotation about parental social life | every 3 days for 6 months
  Visual Analogic scale (1 is unsatisfactory to 10 is satisfactory) quotation about parental social life by participants as assessed by SMARTAUTISM Application V1 2017 (Registered App)
Visual Analogic scale quotation about parental support and resources | every 3 days for 6 months
  Visual Analogic scale (1 is unsatisfactory to 10 is satisfactory) quotation about parental support and resources from third persons by participants as assessed by SMARTAUTISM Application V1 2017 (Registered App)
the duration of use | every 3 days for 6 months
the time of use | every 3 days for 6 months
rate of complete filling | every 3 days for 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Bonnot, PU-PH, Principal Investigator — Nantes CHU
Locations (2):
- France (2):
  - Angers CHU, Angers
  - Nantes CHU, Nantes

REFERENCES:
- [Background] Bonnot O, Bonneau D, Doudard A, Duverger P. Rationale and protocol for using a smartphone application to study autism spectrum disorders: SMARTAUTISM. BMJ Open. 2016 Nov 22;6(11):e012135. doi: 10.1136/bmjopen-2016-012135. PMID 27881525